CLINICAL TRIAL: NCT04325620
Title: A Multicenter, Randomized, Parallel, Double-Blinded, Placebo-controlled Phase 3 Study to Compare Efficacy and Safety of HIP1601 in Patients With Non-Erosive Gastroesophageal Reflux Disease(NERD)
Brief Title: Safety to Evaluate the Efficacy and Safety of HIP1601 in Patients With Non Erosive Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-ESOM-302
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Non-erosive Gastroesphageal Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIP1601 Amg (Experimental): The participants will receive tretment of HIP1601 Amg, orally, once daily for 4weeks.
  Interventions: Drug: HIP1601
- HGP1805 (Placebo Comparator): The participants will receive tretment of HGP1805(Placebo of HIP1601), orally, once daily for 4weeks.
  Interventions: Drug: HGP1805

INTERVENTIONS:
Drug: HIP1601 — HIP1601
  Arms: HIP1601 Amg
Drug: HGP1805 — Placebo of HIP1601
  Arms: HGP1805

SUMMARY:
The purpose of this study is to investigate the safety and clinical efficacy of HIP1601 in patients with Non-erosive gastroesphageal reflux disease.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Parallel, Double-Blinded, Placebo-controlled Phase Ⅲ Study to Compare Efficacy and Safety of HIP1601 in Patients with Non-Erosive Gastroesophageal Reflux Disease(NERD)

ELIGIBILITY:
Inclusion Criteria:

* 19≤ age ≤ 75
* Patients who were not observed mucosal break('not present') according to the LA classification(LA grade) on the EGDEsophago-Gastro-Duodenoscopy
* Patients who had experienced major symptom within 3 months Patients experienced heartburn or acid regurgitation within 7 days of screening day
* Patients who had experienced major symptom within 7 days before randomization. Entry into study also required that patients had experienced at least mild symptoms on at least 2 days/week or at least moderate symptoms on at least 1 day/week based on RDQ
* Patients understood the consents and purpose of this trial and signed consent form

Exclusion Criteria:

* Patients who have erosive GERD, Barrett's esophagus(other significant dysplasia of esophagus), gastroesophageal varicose veins, active peptic ulcer, gastrointestinal bleeding or malignant GI tumor confirmed by endoscopy
* Patients who have a history of gastric or gastroesophageal surgery
* Patients who have Zollinger-Ellison syndrome, eosinophilic esophagitis, primary esophageal motility disorder, acute upper gastrointestinal bleeding, Functional dyspepsia, IBS, IBD within 3 months before Visit 1
* Patients with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary system disease.
* Patients Has a severe liver disorder(AST or ALT level exceeds 3 times more than normal upper range at Visit 1)
* Has a clinically significant renal failure(MDRD eGFR ≤ 59 mL/min/1.73m2 or Serum creatinine >2.0mg/dL at Visit 1)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete resolution of major symptoms at 4-week | 4 week
  Complete resolution is defined as no episodes of symptom during the last 7 days of treatment.

SECONDARY OUTCOMES:
Percentage of patients with complete resolution of major symptoms at 2-week | 2 week
  Complete resolution is defined as no episodes of symptom during the last 7 days of treatment
Frequency and Severity of Reflux disease symptom assessment using Reflux Disease Questionnaire(RDQ) | 2, 4 week
  RDQ frequncy and severity score is 0 to 5 point scale, high score mean a worse outcome.
Time to complete resolution of major symptoms | 4 week
  defined as time to the first day of complete resolution
Resolution rate of major symptoms of first 7 days | 1 week
  defined as first of 7 days with no episodes of symptom using subject's diary
Major symptoms-Free days | 1, 4 week
  Major symptoms-Free days mean rate of days that symtom's severity score is '0' using subject's diary
Quality of Life assessment using Patient Assessment of upper Gastrointestinal disorders-Quality of Life(PAGI-QoL) | 4 week
  PAGI-QoL total score is 0 to 30 point scale, high score mean a better outcome.
Proportion of rescue medication amounts | 4 week
  Use of rescue medication

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No